CLINICAL TRIAL: NCT00000300
Title: Feasibility Study of Take-Home LAAM Medication
Brief Title: Feasibility Study of Take-Home LAAM Medication - 3
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Walter Ling, Principal Investigator, University of California, Los Angeles
Allocation: Randomized | Purpose: Treatment
Other Study IDs: NIDA-09260-3; P50DA009260 (NIH); P50-09260-3
Record Dates: First submitted 1999-09-20; First posted 1999-09-21 (Estimated); Last update posted 2017-11-01 (Actual); Status verified 1995-03

CONDITIONS: Opioid-Related Disorders
Keywords: opiate; dependence
MeSH Terms: conditions — Opioid-Related Disorders | interventions — Methadyl Acetate

INTERVENTIONS:
Drug: LAAM

SUMMARY:
The purpose of this study is to test therapeutic benefits of take-home LAAM. (1) Do subjects with take-home LAAM availability show increased clinical responsibility over subjects without; (2) Do subjects with take-home LAAM attempt diversion when random recall and other diversion safeguards are used; (3) Does treatment response correlate with background or drug use variables at intake, discharge, or during treatment?

DETAILED DESCRIPTION:
1-Year study, participant will be randomly assigned to one of two groups: One will have the opportunity to earn take-home doses by turning in a designated number of clean urines. Two will not have the opportunity to earn take-home doses. Clinic visits three times per week. Urine sample given at each visit.

ELIGIBILITY:
Inclusion Criteria:

meets DSM-IV criteria for opiate dependence. M/F, 18 years or older. Certified for LAAm treatment by a physician. Able to understand english. Willing to provide names, addresses, and numbers of 3 relatives who can aid in patient location for follow-up visits.

Exclusion Criteria:

Hypertensive to LAAM. Pregnant or nursing women. Female of childbearing potential who refuses to use an acceptable form of birth control. Clinically significant abnormality in hematology, blood work, or UA, ETOH and/or sedative/hypnotic dependence according to DSM-IV criteria. Medical or psychiatric illness which would jeopardize safe study participation.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0
Dates: Start 1995-03

PRIMARY OUTCOMES:
Drug use
Retention
Increased prosocial behaviors
Decreased frequency of HIV related behavior

CONTACTS AND LOCATIONS:
Overall Officials: Walter Ling, M.D., Principal Investigator — Friends Research Institute, Inc.
Locations (1):
- Friends Research Institute, Los Angeles, California, United States